CLINICAL TRIAL: NCT00131950
Title: Chicago Breast Health Project, Phase II
Brief Title: Effect of Lifestyle Factors and Hormone Function on Breast Density in Healthy Hispanic Women Who Are Undergoing Mammography for Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: NU-0212-005; CDR0000437805 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2005-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Other: physiologic testing
Other: study of socioeconomic and demographic variables
Procedure: breast imaging study
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Lifestyle factors, such as physical activity, diet, and obesity, and hormone function may affect breast density. Screening tests, such as mammography, may help doctors find tumor cells early and plan better treatment for breast cancer.

PURPOSE: This clinical trial is studying the effect of lifestyle factors and hormone function on breast density in healthy Hispanic women who are undergoing mammography for breast cancer screening.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate physical activity, diet, and obesity, as measured by body mass index and waist circumference, with percent breast density and the absolute estimate of total dense breast area in healthy Hispanic women undergoing screening mammography.
* Correlate fasting serum insulin growth factor (IGF)-1 and the molar ratio of IGF-1 to IGF binding protein-3 with breast density in participants undergoing screening mammography.
* Correlate insulin concentration and insulin resistance with breast density in participants undergoing screening mammography.

OUTLINE: This is a multicenter study.

Participants undergo blood collection and physical examination. Participants also complete breast cancer risk factor, food frequency, and physical activity questionnaires and receive breast health and physical activity education. Participants then undergo a digital screening mammogram. Participants are notified of mammogram results.

PROJECTED ACCRUAL: A total of 114 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy Hispanic women
* Registered patient at the Erie Family Health Centers' West Town or Humboldt Park clinics
* No screening mammography within the past 12 months
* No abnormality on clinical breast exam
* No history of breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 40 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Gapstur, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States